CLINICAL TRIAL: NCT02656212
Title: Early Phase Pre-Clinical and Initial Clinical Research on Epicatechin (Part 2)
Acronym: Epicatechin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency); National Center for Complementary and Integrative Health (NCCIH) (NIH); University of California, San Diego (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Robert R. Henry, MD, Chief, Section of Diabetes, Endocrinology and Metabolism, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08847002; 1R01AT008310-01 (NIH)
Record Dates: First submitted 2016-01-07; First posted 2016-01-14 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Pre-diabetes
Keywords: epicatechin; pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Catechin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (+)-epicatechin 30mg (Experimental): 10 subjects will be randomized to a 30mg dose of synthetic (+)-epicatechin
  Interventions: Drug: epicatechin
- placebo (Placebo Comparator): 5 subjects will be randomized to a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: epicatechin — 30 mg (+)-epicatechin, taken orally, one pill/day in the morning
  Other Names: 122158
  Arms: (+)-epicatechin 30mg
Drug: Placebo — Placebo pill, taken orally, one pill/day in the morning
  Arms: placebo

SUMMARY:
This will be a double-blind, randomized, placebo-controlled, single dose study of (+)- epicatechin with one 30mg dose/day for a total of 7 days

DETAILED DESCRIPTION:
This project is a double-blinded, placebo-controlled, randomized, Phase I study that will include (+)-epicatechin dosing over seven days.

* Subjects will meet the American Diabetes Association (ADA) criteria for pre-diabetes, including impaired fasting glucose (IFG) [refer to inclusion/exclusion criteria].
* The Project includes: 7 day evaluation of a single daily dose of synthetic (+)-epicatechin in pre-diabetic individuals as compared to placebo.
* The Project has 4 outpatient clinic study visits: screening (Visit 1), randomization (Visit 2), end of study drug (Visit 3), follow up end of study (Visit 4).
* This Project has 2 telephone visits

Primary hypothesis: As these studies are designed to evaluate safety and tolerability, there is no primary hypothesis to test.

Primary outcome measures. Vital signs and safety labs: BP, HR, creatinine, alkaline phosphatase, and liver transaminases

These studies will provide initial data about if (+)-epicatechin can influence glycemic control in individuals with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Pre-diabetic based on medical history and screening results
* Male or female
* Must be 21 to 75 years of age (inclusive)
* Able to give informed consent to the procedures
* If female, must be either postmenopausal or test negative for pregnancy at screening and on the day of the procedure. Women on estrogen therapy will be included.
* If female of childbearing potential, must practice and be willing to continue to practice appropriate birth control during the entire duration of the study
* Medication use stable for 4 weeks prior to screening
* Body Mass Index (BMI) > 27 kg/m2
* Definition of pre-diabetes: impaired fasting glucose (IFG, fasting glucose = 100-125 mg/dL) and/OR elevated HbA1c (5.7-6.4%), each in the absence of other risk factors for diabetes

Exclusion Criteria:

* Type 2 diabetes
* Pregnancy
* Younger than 21 or older than 75 years of age
* Clinically significant abnormalities in liver or kidney function (>3x upper limit of normal (ULN)), determined in the last 6 months by a certified clinical laboratory
* Recent myocardial infarct or stroke (within 6 months of screening)
* Blood pressure (BP) >160 mmHg Systolic and >100 mmHg Diastolic
* Medications - thiazolidinediones, any steroids, anti-depressants, weight loss drugs
* Other diseases, besides type 2 diabetes, influencing carbohydrate metabolism

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in major safety endpoints: Blood Pressure (BP) | Baseline and Day 7
  Clinically significant differences in the major safety endpoints are defined as: BP (10 mm Hg change)
Change from baseline in major safety endpoints: Heart Rate (HR) | Baseline and Day 7
  Clinically significant differences in the major safety endpoints are defined as: HR (10 bpm)
Change from baseline in major safety endpoints: Kidney Function | Baseline and Day 7
  Clinically significant differences in the major safety endpoints are defined as: creatinine (>1.5 ULN)
Change from baseline in major safety endpoints: Hepatic Function | Baseline and Day 7
  Clinically significant differences in the major safety endpoints are defined as: highly conservative changes in alkaline phosphatase and liver transaminases (>1.5 ULN)

SECONDARY OUTCOMES:
Change from baseline: Glucose | Baseline and Day 7
  Change from baseline of glucose (mg/dL) as measured from fasting labs collected at Visits 2 and 3.
Change from baseline: Insulin | Baseline and Day 7
  Change from baseline of insulin (uIU/ml) as measured from fasting labs collected at Visits 2 and 3.
Change from baseline: C-Peptide | Baseline and Day 7
  Change from baseline of C-Peptide (ng/mL) as measured from fasting labs collected at Visits 2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Henry, MD, Principal Investigator — San Diego Veterans Healthcare System
Locations (2):
- United States (2):
  - CMR Center for Metabolic Research VASDHS, San Diego, California
  - VA San Diego Healthcare System, San Diego, California